CLINICAL TRIAL: NCT02138994
Title: Clinical Assessment of the Next Science Wound Gel Efficacy in Chronic Wound Compared to Standard of Care
Brief Title: Next Science Wound Gel Efficacy in Chronic Wound Versus Standard of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Next Science TM (Industry)
Collaborators: Mayo Clinic (Other); Jacksonville Center For Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP-001
Record Dates: First submitted 2014-05-12; First posted 2014-05-15 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Wound Chronic Draining

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triple Antibiotic Ointment Neosporin (Active Comparator): Daily direct application to the wound, covered with conventional dressing. Dressing should be changed daily or as directed by the health care provider.
  Interventions: Drug: Triple Antibiotic Ointment Neosporin
- Next Science Wound Gel (Experimental): Daily direct application to the wound, covered with a conventional non-alginate dressing. Dressing should be changed daily or as directed by the health care provider.
  Interventions: Device: Next Science Wound Gel

INTERVENTIONS:
Device: Next Science Wound Gel
  Arms: Next Science Wound Gel
Drug: Triple Antibiotic Ointment Neosporin — Subjects randomized to Neosporin will be required to complete 1 month of treatment comprising a screening/baseline, 2-week and 1-month visits. After 1 month the following may occur based on wound progression and/or the investigator's clinical judgment:
  * Subject may continue the application of Neosporin until wound closure or
  * Subject may cross over to the treatment group for 3 months
  Arms: Triple Antibiotic Ointment Neosporin

SUMMARY:
This is a 3 to 4 months, multi-site, prospective randomized clinical study of patients diagnosed with a chronic wound. The primary objective is to assess changes in healing rate, by measuring differences in wound area when treating chronic wounds with the Next Science Wound Gel compared to the Triple Antibiotic Ointment Neosporin (Standard of Care, SOC). At the end of the study period, patients may continue receiving their assigned study treatment provided they have signed the "Continuation of Treatment Informed Consent" and the rational for continuation is documented by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older
* Presence of full-thickness wound for more than one month (i.e. chronic)
* Ulcer must be greater than 1 centimeter in area to enable biofilm sampling
* NOT a candidate for vascular reconstructive surgery to restore blood flow to the wound
* Willing to comply with all study procedures and be available for the duration of the study
* Provide signed and dated informed consent

Exclusion Criteria:

* Subjects unable to provide signed and dated informed consent
* Male or female less than 18 years old
* Presence of a full-thickness wound for less than one month
* A candidate for vascular reconstructive surgery to restore blood flow to the wound
* Subjects with bleeding dyscrasia or with medical conditions that would make a bleeding complication likely
* Subjects who's wound is less than 1 cm precluding adequate wound biofilm sampling
* Subject with known allergic reaction to the study products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Wound Size Reduction | 2, 4, 8 and 12 weeks

SECONDARY OUTCOMES:
Wound Closure | 2, 4, 8 and 12 weeks

OTHER OUTCOMES:
Reduction of bacterial species types and amounts | 0 and 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Jacksonville Center for Clinical Research - RCCR location, Jacksonville, Florida